CLINICAL TRIAL: NCT02487069
Title: Allogeneic Stem Cell Transplantation With Alternative Donor in Treatment of Hematologic Malignancy
Brief Title: Allo-HSCT With Alternative Donor in Treatment of Hematologic Malignancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Guangzhou First People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Zhujiang Hospital (Other); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Fujian Medical University Union Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alternative Donor HSCT-2015
Record Dates: First submitted 2015-06-14; First posted 2015-07-01 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2019-03

CONDITIONS: Acute Leukemia; Chronic Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes | interventions — Cyclosporine; Methotrexate; Antilymphocyte Serum; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MSD group (Experimental): The patients will received HSCT from MSD.
  Interventions: Procedure: HSCT from MSD; Drug: Cyclosporin A; Drug: Methotrexate; Drug: Mycophenolate mofetil
- MUD group (Experimental): The patients will received HSCT from MUD.
  Interventions: Procedure: HSCT from MUD; Drug: Cyclosporin A; Drug: Methotrexate; Drug: Antithymocyte globulin
- HRD group (Experimental): The patients will received HSCT from HRD.
  Interventions: Procedure: HSCT from HRD; Drug: Cyclosporin A; Drug: Methotrexate; Drug: Antithymocyte globulin; Drug: Mycophenolate mofetil

INTERVENTIONS:
Procedure: HSCT from MSD — HSCT from MSD is the first choice for the patients who have HLA-matched sibling donors.
  Arms: MSD group
Procedure: HSCT from MUD — HSCT from MUD is the second choice for the patients who don't have HLA-matched sibling donors but have HLA-matched unrelated donors.
  Arms: MUD group
Procedure: HSCT from HRD — HSCT from HRD is the choice for the patients who have neither HLA-matched sibling donors nor HLA-matched unrelated donors.
  Arms: HRD group
Drug: Cyclosporin A — CsA is used in all the patients for GVHD prophylaxis.
  Other Names: CsA
Drug: Methotrexate — MTX is used in all the patients for GVHD prophylaxis.
  Other Names: MTX
Drug: Antithymocyte globulin — ATG is used in the patients receiving HSCT from MUD and HRD for GVHD prophylaxis.In MUD group,total ATG doses is 7 mg/kg;In HRD group,total ATG doses is 7.5 or 10 mg/kg.
  Other Names: ATG
  Arms: HRD group; MUD group
Drug: Mycophenolate mofetil — MMF is used in the patients receiving HSCT from MSD and HRD for GVHD prophylaxis.
  Other Names: MMF
  Arms: HRD group; MSD group

SUMMARY:
The purpose of this study is to compare the efficacy of allogeneic hematopoietic stem cell transplantation (allo-HSCT) from matched sibling donor (MSD),matched unrelated donor (MUD) and haploidentical related donors(HRD) in the treatment of hematologic malignancy.

DETAILED DESCRIPTION:
Currently, allogeneic hematopoietic stem cell transplantation (allo-HSCT) remains the only curative therapy for a majority of malignant hematologic diseases, especially acute leukemia. HSCT from MSD offers the best results for these diseases, but lack of this donor resource has restricted its wide application. HSCT from MUD provides another option, but MUDs still cannot satisfy all patients due to unsuccessful donor searches. Almost all patients have an available related donor with whom they share a single HLA haplotype (ie, haploidentical related donor), and it owns the advantage of immediate availability, especially for those who urgently need transplantation.The results of transplantation from HRD have improved significantly over the past few years. However, the results from such haploidentical transplantation have not formally been compared with those of transplantation in patients contemporaneously using MSDs and MUDs for hematologic malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary disease is acute leukemia/MDS/CML
* Receiving allo-HSCT

Exclusion Criteria:

* cardiac dysfunction (particularly congestive heart failure)
* hepatic abnormalities (bilirubin ≥ 3 mg/dL, aminotransferase> 2 times the upper limit of normal)
* renal dysfunction (creatinine clearance rate < 30 mL/min)
* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 876 (Actual)
Dates: Start 2015-06; Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 year
  The primary endpoint is overall survival within 3 years after HSCT.

SECONDARY OUTCOMES:
Disease-free survival | 3 year
Incidence of transplantation-related mortality | 3 year
Incidence of graft-versus-host disease | 3 year
  Graft-versus-host disease include acute and chronic Graft-versus-host disease
Incidence of infection | 3 year
  Infection includes bacterial, fungal and viral infections.
hematopoietic reconstruction | 1 year
  Hematopoietic reconstruction includes the time of neutrophil and platelet reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Luo Y, Xiao H, Lai X, Shi J, Tan Y, He J, Xie W, Zheng W, Zhu Y, Ye X, Yu X, Cai Z, Lin M, Huang H. T-cell-replete haploidentical HSCT with low-dose anti-T-lymphocyte globulin compared with matched sibling HSCT and unrelated HSCT. Blood. 2014 Oct 23;124(17):2735-43. doi: 10.1182/blood-2014-04-571570. Epub 2014 Sep 11. PMID 25214441
- [Background] Lu DP, Dong L, Wu T, Huang XJ, Zhang MJ, Han W, Chen H, Liu DH, Gao ZY, Chen YH, Xu LP, Zhang YC, Ren HY, Li D, Liu KY. Conditioning including antithymocyte globulin followed by unmanipulated HLA-mismatched/haploidentical blood and marrow transplantation can achieve comparable outcomes with HLA-identical sibling transplantation. Blood. 2006 Apr 15;107(8):3065-73. doi: 10.1182/blood-2005-05-2146. Epub 2005 Dec 27. PMID 16380454
- [Derived] Ling Y, Xuan L, Xu N, Huang F, Fan Z, Guo Z, Xu X, Liu H, Lin R, Yu S, Zhang H, Jin H, Wu M, Liu C, Liang X, Ou R, Zhang Y, Liu X, Qu H, Zhai X, Sun J, Zhao Y, Liu Q. Busulfan Plus Fludarabine Compared With Busulfan Plus Cyclophosphamide for AML Undergoing HLA-Haploidentical Hematopoietic Cell Transplantation: A Multicenter Randomized Phase III Trial. J Clin Oncol. 2023 Oct 10;41(29):4632-4642. doi: 10.1200/JCO.23.00101. Epub 2023 Jun 19. PMID 37335960